CLINICAL TRIAL: NCT04317846
Title: TransRadIal Evaluation STudy of diamEter Increase After Vasodilatory Drugs Administration: The TRIESTE Randomized Study
Brief Title: Transradial Evaluation Study of Diameter Increase After Vasodilatory Drugs Administration.
Acronym: TRIESTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Centre de recherche clinique - FBM-CHUV (Unknown)
Responsible Party: Principal Investigator, Vladimir Rubimbura, Principal Investigator, Dr Vladimir Rubimbura, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Trieste-study
Record Dates: First submitted 2020-03-18; First posted 2020-03-23 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Arterial Spasm; Coronary Artery Disease
Keywords: radial spasm; percutaneous coronary intervention; vasodilatory drugs
MeSH Terms: conditions — Coronary Artery Disease; Spasm

STUDY DESIGN:
Intervention Model Description: Multi-center randomised controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intra-radial group (Active Comparator): intra-radial administration of the vasodilatory drugs after sheath insertion (verapamil 2.5 mg + isosorbide dinitrate 0.5 mg)
  Interventions: Other: Intravenous administration of vasodilatory drugs
- Intravenous-post group (Experimental): intra-venous administration of the vasodilatory drugs after sheath insertion (verapamil 2.5 mg + isosorbide dinitrate 0.5 mg)
  Interventions: Other: Intravenous administration of vasodilatory drugs
- Intravenous-pre group (Experimental): intra-venous administration of the vasodilatory drugs 5 minutes before sheath insertion (verapamil 2.5 mg + isosorbide dinitrate 0.5 mg)
  Interventions: Other: Intravenous administration of vasodilatory drugs

INTERVENTIONS:
Other: Intravenous administration of vasodilatory drugs — Administration of the vasodilatory drugs in a different pattern than intra-arterially

SUMMARY:
Radial artery access use in percutaneous cardiac interventions (PCI) is associated with a lower risk of vascular complications, bleeding and major adverse cardiac events including cardiac death in the long-term follow-up. Intra-radial administration of vasodilatory drugs, transiently painful for the patient, reduces the risk of spasm and is currently the standard technique performed worldwide. However, the efficacy of intravenous administration of vasodilatory drugs has never been evaluated.

DETAILED DESCRIPTION:
Multicenter, randomised controlled trial, designed to evaluate the noninferiority of the intravenous administration of vasodilatory drugs in comparison with the actual gold standard intra-arterial radial route, in terms of radial artery diameter increase.

All consecutive patients with stable ischemic disease or stable acute coronary syndrome (NSTEMI - Non-ST elevation myocardial infarction) for whom a coronary procedure is planned will be included in the study. Three groups will be constituted. For all groups, the diameters of both radial arteries will be measured thrice by echo-Doppler: 5 minutes before sheath insertion, immediately before sheath insertion and 5 minutes after sheath insertion. Pain evaluation will be performed after injection of the vasodilatory drugs/placebo in the radial artery:

* Group 1 (control group): intra-radial administration of the vasodilatory drugs after sheath insertion (verapamil 2.5 mg + isosorbide dinitrate 0.5 mg)
* Group 2 (intravenous-post): intra-venous administration of the vasodilatory drugs after sheath insertion (verapamil 2.5 mg + isosorbide dinitrate 0.5 mg)
* Group 3 (intravenous-pre): intra-venous administration of the vasodilatory drugs 5 minutes before sheath insertion (verapamil 2.5 mg + isosorbide dinitrate 0.5 mg)

ELIGIBILITY:
Inclusion criteria:

1. Clinical indication for a coronary angiogram by radial route
2. Age ≥18 years old
3. Chronic coronary disease or stable acute coronary syndrome (NSTEMI, Non-ST Elevation Myocardial Infarction)

Exclusion criteria:

1. ST-Elevation Myocardial infarction
2. Severe aortic stenosis (aortic valve area <0.8 cm2 or mean gradient > 40 mmHg)
3. Severe left ventricular dysfunction (left ventricular ejection fraction < 30%).
4. Heart failure, hemodynamic instability or severe hypotension (systolic arterial pressure < 90 mm Hg or heart rate < 45 bpm).
5. Atrioventricular disturbances (atrioventricular block 2° or 3°).
6. Contraindications to the class of drugs used in the trial, e.g. known hypersensitivity or allergy to class of drugs or the investigational
7. Women who are pregnant or breast feeding, Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
8. Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
9. Psychological disorders, dementia, etc. of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Maximal radial artery diameter dilation, measured by echo-doppler, after administration of vasodilatory drugs by intravenous or intra-radial route. | 5 minutes after vasodilatory drugs administration
  Radial artery diameter

SECONDARY OUTCOMES:
Pain evaluation after vasodilatory drugs administration using the intravenous versus intra-radial route | Procedure (During vasodilatory drugs administration)
  Scale from 0 to 10, lower values corresponding to lower pain and higher values to intense pain.
Hemodynamic changes after vasodilatory drugs administration using the intravenous versus intra-radial route | 5 minutes after vasodilatory drugs administration
  Measure of arterial pressure
Heart rate change after vasodilatory drugs administration using the intravenous versus intra-radial route | 5 minutes after vasodilatory drugs administration
  Measure of heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Rubimbura, MD, Principal Investigator — MD
Locations (2):
- Switzerland (2):
  - Rubimbura Vladimir, Lausanne, Canton of Vaud
  - Morges Hospital, Morges, Canton of Vaud

IPD SHARING:
Plan to Share IPD: No